CLINICAL TRIAL: NCT02712684
Title: Multi-parametric Ultrasound Targeted Biopsies Compared to Multi-parametric MRI Targeted Biopsies in the Diagnosis of Clinically Significant Prostate Cancer
Brief Title: Cancer Diagnosis by Multiparametric UltraSound of the Prostate
Acronym: CADMUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0473
Record Dates: First submitted 2016-02-04; First posted 2016-03-18 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: multiparametric MRI. Multi-parametric ultrasound — The investigators aim to test the hypothesis that multiparametric ultrasound is able to detect clinically significant prostate cancer with an accuracy that is similar to multiparametric MRI. Multi-parametric ultrasound uses different types of ultrasound images to visualise different aspects of the tissue. In other words, the standard grey-scale images shows the gross anatomy, Power Doppler and Contrast enhanced Ultrasound image blood supply (cancers have more blood supply), and Real-Time Elastography images the density of tissue (cancers are more dense).

SUMMARY:
In men who require a prostate biopsy does a multi-parametric ultrasound based diagnostic strategy compared to a multi-parametric MRI based diagnostic strategy lead to similar detection of clinically significant prostate cancer?

DETAILED DESCRIPTION:
Men who require prostate biopsy will be approached and consented to enter this study. Participants will all undergo pre-biopsy mp-MRI and mp-USS of the prostate. Only men with positive scans will undergo prostate biopsy. The order in which lesions discovered on mp-MRI or on mp-USS are sampled will be randomised. All biopsies will be taken via the transperineal route in a single procedure. Comparison will be drawn between biopsy results of lesions detected by mp-USS with those lesions detected by mp-MRI. Consideration will be given as to whether a lesion detected by one imaging modality is the same abnormality as one detected by the other imaging modality, in the same patient. Analysis will be carried out at both the level of the lesion and the whole prostate. Men without suspicious lesions on either imaging modality will not proceed to biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. A potential need for prostate biopsy indicated by raised PSA or other clinical parameter, the final decision over which will be taken after imaging.
2. PSA </=20ng/ml measured within 6 months of screening visit
3. An understanding of the English language sufficient to understand written and verbal information about the trial and consent process
4. Estimated life expectancy of 5 years or more
5. Signed informed consent

Exclusion Criteria:

1. Any contraindication to the ultrasound contrast agent including right to left shunt, pulmonary hypertension, uncontrolled hypertension and adult respiratory distress syndrome. Also patients with a recent acute coronary syndrome or unstable ischaemic heart disease.
2. Any form of hormones (except 5-alpha reductase inhibitors) within 6 months of screening visit
3. Irreversible coagulopathy predisposing to bleeding
4. Inability to undergo transrectal ultrasonography
5. Prostate volume, measured at the time of mp-USS if previously unknown, of >60cc.
6. Previous radiation therapy to the prostate
7. Previous HIFU, cryosurgery, thermal therapy, irreversible electroporation, photodynamic, photothermal therapy, microwave or injectable toxin therapy to the prostate.
8. Transurethral resection or vaporization of the prostate for benign prostatic hyperplasia using any energy modality within 6 months of screening visit
9. Nodal or metastatic prostate cancer on any form of imaging at any time-point
10. Not fit for general anaesthetic
11. Any other condition the investigator considers would make the patient unsuitable

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men at or referred to the participating centres who may require a prostate biopsy. Referrals will be screened and potential participants contacted by telephone, post or email. These men will be given the patient information sheet at least 24 hours before their clinic visit, allowing adequate time to consider their desire for involvement
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
To determine the overall agreement in identifying lesions to biopsy between mp-USS and mp-MRI in men who require a prostate biopsy. Then compare agreement in proportion of men diagnosed with clinically significant prostate cancer on biopsy. | at time of surgery
  Clinically significant for the purpose will be defined by UCL/Ahmed definition 1:Gleason ≥4+3 and/or maximum cancer core length of ≥ 6mm

SECONDARY OUTCOMES:
To compare the overall agreement in proportion of men diagnosed with other thresholds of clinically significant prostate cancer on biopsy | at time of surgery
  Thresholds for clinical significance namely UCL/Ahmed definition 2 (a) Gleason ≥ 3+4 and/or Maximum cancer core length ≥ 4mm, (b) Gleason ≥ 3+4 and or MCCL ≥ 6mm (c) Any length of Gleason ≥ 3+4 (d) Any length of Gleason ≥4+3
To determine the detection of clinically significant cancer (using all of the pre-specified definitions based on histology) by using the combination of these two imaging techniques versus either modality alone | at time of surgery
To determine whether the order in which the targeted biopsies are carried out, either to the same target (present on both scans) or different targets impacts on detection of clinically significant cancer | at time of surgery
  clinically significant cancer (using all of the pre-specified definitions based on histology)
To compare, in those men who go on to radical prostatectomy, the mp-MRI, mp-USS and histology from targeted biopsy with the whole mount specimen obtained at surgery. | at time of surgery
To create an inception cohort of men, consented for long-term follow-up and linkage, providing the potential for further translational and clinical studies | at time of surgery
To determine rates of adverse events, resource utilization and impact of each test on health-related quality-of-life (using EQ-5D-5L questionnaire) which would allow modelling of overall cost-effectiveness of one strategy compared to the other. | at time of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospitals, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Velonas VM, Woo HH, dos Remedios CG, Assinder SJ. Current status of biomarkers for prostate cancer. Int J Mol Sci. 2013 May 24;14(6):11034-60. doi: 10.3390/ijms140611034. PMID 23708103
- [Result] Kirkham AP, Haslam P, Keanie JY, McCafferty I, Padhani AR, Punwani S, Richenberg J, Rottenberg G, Sohaib A, Thompson P, Turnbull LW, Kurban L, Sahdev A, Clements R, Carey BM, Allen C. Prostate MRI: who, when, and how? Report from a UK consensus meeting. Clin Radiol. 2013 Oct;68(10):1016-23. doi: 10.1016/j.crad.2013.03.030. Epub 2013 Jul 1. PMID 23827086
- [Result] Welch HG, Albertsen PC. Prostate cancer diagnosis and treatment after the introduction of prostate-specific antigen screening: 1986-2005. J Natl Cancer Inst. 2009 Oct 7;101(19):1325-9. doi: 10.1093/jnci/djp278. Epub 2009 Aug 31. PMID 19720969
- [Result] Wilt TJ, Ahmed HU. Prostate cancer screening and the management of clinically localized disease. BMJ. 2013 Jan 29;346:f325. doi: 10.1136/bmj.f325. No abstract available. PMID 23360718
- [Result] Wei JT. Limitations of a contemporary prostate biopsy: the blind march forward. Urol Oncol. 2010 Sep-Oct;28(5):546-9. doi: 10.1016/j.urolonc.2009.12.022. PMID 20816614
- [Result] Thompson IM, Ankerst DP, Tangen CM. Prostate-specific antigen, risk factors, and prostate cancer: confounders nestled in an enigma. J Natl Cancer Inst. 2010 Sep 8;102(17):1299-301. doi: 10.1093/jnci/djq313. Epub 2010 Aug 19. No abstract available. PMID 20724727
- [Derived] Grey ADR, Scott R, Shah B, Acher P, Liyanage S, Pavlou M, Omar R, Chinegwundoh F, Patki P, Shah TT, Hamid S, Ghei M, Gilbert K, Campbell D, Brew-Graves C, Arumainayagam N, Chapman A, McLeavy L, Karatziou A, Alsaadi Z, Collins T, Freeman A, Eldred-Evans D, Bertoncelli-Tanaka M, Tam H, Ramachandran N, Madaan S, Winkler M, Arya M, Emberton M, Ahmed HU. Multiparametric ultrasound versus multiparametric MRI to diagnose prostate cancer (CADMUS): a prospective, multicentre, paired-cohort, confirmatory study. Lancet Oncol. 2022 Mar;23(3):428-438. doi: 10.1016/S1470-2045(22)00016-X. PMID 35240084